CLINICAL TRIAL: NCT03214913
Title: Controlled Fluid Resuscitation Strategy in Sepsis Patient
Brief Title: Controlled Fluid Resuscitation in Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Erzhen Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sepsis Fluid 1
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Sepsis
Keywords: resuscitation; fluid therapy
MeSH Terms: conditions — Sepsis | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGDT Group (Other): Early Goal Directed Therapy ：30ml/kg in the first bolus to have a CVP（central venous pressure） 8-12 mmHg and MAP（mean artery pressure ） 65-85 mm Hg,and urine output ≥0.5 ml/kg/h, ScvO2 ≤70%；If not, use noradrenaline，red blood cell transfusion if necessary.
  Interventions: Other: Early Goal Directed Therapy
- Ruijin Group (Other): Ruijin Strategy therapy：10~5ml/kg/h，crystalloid vs colloid 2:1 resuscitation;using noradrenaline at the same time;red blood cell transfusion if necessary.
  target： fulfillment of two or more of four criteria:1. HR（heart rate） <120 beats/min, 2.MAP 65-85 mm Hg, 3. urine output ≥1 ml/kg /h 4. HCT（hematocrit） 25%~35%.
  Interventions: Other: Ruijin Strategy

INTERVENTIONS:
Other: Early Goal Directed Therapy — EGDT therapy ：30ml/kg in the first bolus to have a CVP 8-12 mmHg and MAP 65-85 mm Hg,and urine output ≥0.5 ml/kg/h, ScvO2 ≤70%；If not, use noradrenine，red blood cell transfusion if necessary.
  Other Names: EGDT therapy
  Arms: EGDT Group
Other: Ruijin Strategy — Ruijin Strategy：10~5ml/kg/h，crystalloid vs colloid 2:1 resuscitation;using noradrenaline at the same time;red blood cell transfusion if necessary.
  target： fulfillment of two or more of four criteria:1. HR <120 beats/min, 2.MAP 65-85 mm Hg, 3. urine output ≥1 ml/kg /h 4. HCT 25%~35%.
  Other Names: controlled fluid therapy
  Arms: Ruijin Group

SUMMARY:
To evaluate two different strategy of fluid resuscitation in sepsis patients

DETAILED DESCRIPTION:
Early goal-directed fluid therapy (EGDT) had been regarded as an important fluid therapy strategy in early sepsis or septic shock patients. In recent years, several randomized control studies showed the EGDT therapy cannot make a better outcome in sepsis patients compared to the standard therapy. A strategy of controlled fluid resuscitation had showed good outcome in critical illness such as severe acute pancreatitis, major trauma. But many aspects of the so-called controlled fluid resuscitation remained controversial. In a previous study on severe acute pancreatitis, we described a bundle of controlled fluid resuscitation which had showed an ideal result with higher survival rate. So, we are going to use the bundle on sepsis patients, and to see if it can bring a better out come in sepsis patients compared to the EGDT strategy. This study aims to determine a better strategy of fluid resuscitation in sepsis patients

ELIGIBILITY:
Inclusion Criteria:

* 1.sepsis patients in accordance with the Sepsis 3.0 definition(SOFA increase ≥2 compared to the baseline，due to infection )
* 2.the first blood lactate in our hospital is ≥ 4mmol/L or MAP<90mmHg after 20ml/kg fluid bolus
* 3.the shock is diagnosed within 24hrs after onset

Exclusion Criteria:

* - 1.<18 years old
* 2.Pregnancy
* 3 with co-morbidity such as AE-COPD, stroke, seizure, lung edema, acute coronary syndrome
* 4 with contra-indication of CVC(central venous catheter) placement
* 5 trauma or major burn
* 6 poisoning
* 7 any cancer receiving chemotherapy
* 8.immunosuppression (for organ transplantation or disease of immune system)
* 9.acute pancreatitis
* 10.relapse sepsis

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | the 28th day from enrolled
  Mortality

SECONDARY OUTCOMES:
Mortality | the 60th day from enrolled
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Er Chen, Study Director — Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao EQ, Tang YQ, Fei J, Qin S, Wu J, Li L, Min D, Zhang SD. Fluid therapy for severe acute pancreatitis in acute response stage. Chin Med J (Engl). 2009 Jan 20;122(2):169-73. PMID 19187641
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338